CLINICAL TRIAL: NCT04733625
Title: The Effect of Vitamin D Therapy on Morbidity and Moratlity in Patients With SARS-CoV 2 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA-2020/151
Record Dates: First submitted 2021-01-31; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention(Vitamin D therapy (Active Comparator): 40 patients with diabetes and vitamin D deficinecy that are Covid-19 positive. a single dose of Cholecaciferol will be administered
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): 16 diabetic patients with vitamin D deficiancy and COVID-19 POSITIVE
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — single injection of Vitamin D (200000 I.U
  Other Names: vitamin D
  Arms: Intervention(Vitamin D therapy
Drug: Placebo — placebo medication
  Arms: Placebo

SUMMARY:
The ongoing pandemic of SARS CoV-2 virus is calling for effective preventive and theraputic interventions. Vitamin D has been shown to play immunemodulatory functions in human. Low vitamin D levels have been linked to increased susciptability to infections especially the acute respiratory infections. This randomised controlled study aims to explore the effect of vitamin D administration on the outcome of SARS- CoV2 virus

DETAILED DESCRIPTION:
Background: Coronavirus disease COVID-19 is an ongoing pandemic and is causing avoidable fatalities worldwide. Vitamin D plays an essential role in the immune system. Vitamin D interferes with the majority of the immune systems cells such as macrophages, B and T lymphocytes, neutrophils and dendritic cells. We aim to find whether supplementation of vitamin D deficient diabetes with a single intramuscular cholecalciferol injection could improve the prognosis of those patients.

Patients and Methods: This was a placebo controlled randomized prospective study, included cohorts of 40 diabetes elderly patients who got infected with SARS-CoV-2 compared with 16 elderly diabetes patients matched of the same age group who got infected with SARS-CoV-2 but given a placebo instead intramuscularly were used as a control. Clinical, laboratory, treatment, and outcome data were recorded after six weeks of follow up especially ICU admissions and fate of COVID-19 disease.Vitamin D was given as a single intramuscular injection during period of the study.

ELIGIBILITY:
Inclusion Criteria:

- Elderly type II diabetes adult with age more than 60 years males and females having deficient serum vitamin D levels (less than 25 ng/ml).

Diabetes patients recruited to the control group were only included in the study if not known to have cholecalciferol supplementation within last 6 weeks. All elderly vitamin D deficient diabetes patients were diagnosed with COVID-19 when throat-swab specimens for SARS-CoV-2 PCR were positive.

Exclusion Criteria:

* patients with known history of renal stones, diagnosis of hypercalcemia with the past year, baseline serum total calcium more than 10mg/dl, established diagnosis associated with increase the risk of hypercalcemia (e.g. metastatic cancer, sarcoidosis, multiple myeloma, primary hyperparathyroidism), and current vitamin D supplementation

Moreover, other exclusion criteria included those with known malignancy, with organ transplant, and those with known chronic autoimmune diseases and lastly those on systemic steroid for any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Death or need for intubation | 6 weeks
  In hospital death or need for intubation

CONTACTS AND LOCATIONS:
Overall Officials: Amin Roshdy, PHD, Principal Investigator — Kasr Alainy faculty of medicine
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No